CLINICAL TRIAL: NCT00219362
Title: A Phase II, Randomized, Placebo-controlled Study to Evaluate the Immunogenicity and the Safety of 2 Schedules of an Homologous Prime-boost With the ALVAC-HIV vCP1452 in Chronically HIV-Infected Patients
Brief Title: Immunogenicity and Safety of 2 Schedules of ALVAC-HIV vCP1452 in Chronically HIV-Infected Patients
Acronym: MANON 02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Objectif Recherche Vaccins SIDA (Other)
Responsible Party: Pr Christine KATLAMA, Objectif Recherche Vaccins SIDA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORVACS 002
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infection
Keywords: HIV-1 infection; therapeutic vaccine; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — N-(8-aminohexyl)-5-iodonaphthalene-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ALVAC-HIV 4 injections (Experimental): Arm A: injection of ALVAC-HIV(vCP1452) for a total of 4 injections (W0, W4, W8, W20)
  Interventions: Biological: one injection of vCP1452 at W0, W4, W8 and W20
- ALVAC-HIV 3 injections (Experimental): Arm B: injection of ALVAC-HIV(vCP1452) for a total of injections (W4, W8, W20)
  Interventions: Biological: one injection of vCP1452 at W4, W8 and W20
- Placebo - 4 injections (Placebo Comparator): Arm C1: injection of placebo for a total of 4 injections (W0, W4, W8, W20)
  Interventions: Biological: one injection of placebo at W0, W4, W8, W20 or at W4, W8,W20
- Placebo - 3 injections (Placebo Comparator): Arm C2: injection of placebo for a total of 3 injections (W4, W8, W20)
  Interventions: Biological: one injection of placebo at W0, W4, W8, W20 or at W4, W8,W20

INTERVENTIONS:
Biological: one injection of vCP1452 at W0, W4, W8 and W20
  Arms: ALVAC-HIV 4 injections
Biological: one injection of vCP1452 at W4, W8 and W20
  Arms: ALVAC-HIV 3 injections
Biological: one injection of placebo at W0, W4, W8, W20 or at W4, W8,W20
  Arms: Placebo - 3 injections; Placebo - 4 injections

SUMMARY:
Prior pilot studies have shown that four monthly injections of ALVAC-HIV (vCP1433) are immunogenic in 60% HIV-infected patients with a boosting effect obtained after 1 or 2 injections followed by a plateau or a decrease of these responses prior to interrupting therapy. The goal of the present study is to look for an improved vaccination schedule in terms of strength and duration of the HIV-specific immunity induced by the HIV-recombinant canary pox vector ALVAC-HIV (vCP1452) by testing a strategy of immunization involving a first series of two versus three monthly injections followed by a boost three months later.

DETAILED DESCRIPTION:
Manon 02 is a phase II, multicentre, randomized, placebo-controlled study with 3 arms comprising 2 steps:

Step I : Immunization phase from W0 to W24, on HAART

The immunization will be administered by intramuscular injection :

Arm A: one injection of vCP1452 at W0, W4, W8 and W20 + HAART, for a total of 4 injections Arm B: one injection of vCP1452 at W4, W8 and W20 + HAART, for a total of 3 injections Arm C: one injection of placebo at W0, W4, W8 and W20 + HAART, for a total of 4 injections or at W4, W8 and W20 + HAART, for a total of 3 injections

Step II: Post immunization phase from W24 to W48, off HAART

Discontinuation of antiretroviral therapy (ARV) from W24 to W48 :

The ARV treatment interruption will be proposed at W24, 4 weeks after the last immunization, to patient who had completed their immunization phase and have CD4 cell counts > 350 cells/mm3 and HIV plasma RNA < 400 cp/ml.

In order to be able to evaluate the capacity of the immune response to reduce the viral replication, a period of 16 weeks of interruption is recommended from W24 to W40.

Resumption of antiretroviral therapy :

From W24 to W40 : During this 16 weeks period, in case of a decline of CD4 cell counts below 250 cells/mm3 or of a loss of CD4 greater than 50% of the baseline value, HAART will be restarted.

From W40 to W48 : HAART should be reintroduced if HIV-1 RNA levels > 50 000 cp/ml on 2 consecutive measurements at two weeks interval even if the CD4 counts are above 250 cells/mm3.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* under potent antiretroviral therapy for more than 6 months
* with entry CD4+ counts > 350 cells/mm3 for at least 1 year
* plasma HIV RNA < 400 cp/ml for at least the last 6 months
* Contraception needed for women

Exclusion Criteria:

* Antiretroviral therapy started with CD4 cell count > 400/mm3
* Patients treated at time of primary HIV infection
* Patient with past AIDS defining event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-04; Primary Completion 2005-11 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the frequency of HIV-specific PBMC (CD4/CD8) at W24 (4 weeks after the last immunization)

SECONDARY OUTCOMES:
- Percentage of responders as defined by an increase of at least 0.7 log10 from baseline of the frequencies of HIV-specific PBMC and/or CD4 and/or CD8 T cells four weeks after the last immunization(W24) as measured by ELISpot IFNγ
- Change from baseline of the frequency of HIV-specific PBMC and/or CD4 and/or CD8 T cells at week 4, 6, 8, 12, 20 and 24 in the study arms as measured by ELISpot IFNγ
- Evaluation of the magnitude of CD4 and CD8 T cell response at W4, W6, W8, W12, W20, W24 in the study arms
- Evaluation of the immune responses, HIV-specific PBMC and/or CD4 and/or CD8 T cells at W48
- Percentage of patients who generate a primary immune response against the artificial pol/nef sequences present in the vaccine but not in the HIV strain
- Evaluation of the immune responses directed to vCP1452 in the study arms at all study point during the immunization phase
- Percentage of patients who do not reach the restart therapy criteria from W24 to W48
- Percentage of patients who remain off therapy at W48
- Evaluation of the safety and tolerability of the vCP1452

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Study Chair — Services des maladies infectieuses et tropicales, Hopital de la Pitié-Salpétrière, Université Pierre et Marie Curie, INSERM U720
Locations (5):
- Northwestern University Medical School, Chicago, Illinois, United States
- Service des maladies infectieuses et tropicales, Hopital Pitié-Salpétrière, Pavillon Laveran, Paris, France
- Klinikum der Johann Nolfgang Goethe Universitat Zentrum des Innerin Medizin, Frankfurt am Main, Germany
- Spain (2):
  - Fundacio Irsi Caixa Retrovirology Laboratory, Hospital Universitari Germans, Badalona
  - Servicios de Infecciosos, Hospital y clinic Provincial, Barcelona

REFERENCES:
- [Background] Autran B, Debre P, Walker B, Katlama C. Therapeutic vaccines against HIV need international partnerships. Nat Rev Immunol. 2003 Jun;3(6):503-8. doi: 10.1038/nri1107. PMID 12776210
- [Background] Autran B, Costagliola D, Murphy R, Katlama C. Evaluating therapeutic vaccines in patients infected with HIV. Expert Rev Vaccines. 2004 Aug;3(4 Suppl):S169-77. doi: 10.1586/14760584.3.4.s169. PMID 15285715
- [Result] Autran B, Murphy RL, Costagliola D, Tubiana R, Clotet B, Gatell J, Staszewski S, Wincker N, Assoumou L, El-Habib R, Calvez V, Walker B, Katlama C; ORVACS Study Group. Greater viral rebound and reduced time to resume antiretroviral therapy after therapeutic immunization with the ALVAC-HIV vaccine (vCP1452). AIDS. 2008 Jul 11;22(11):1313-22. doi: 10.1097/QAD.0b013e3282fdce94. PMID 18580611